CLINICAL TRIAL: NCT01965574
Title: Evaluation of Performance Diagnosis of Hemodynamic Parameters of Preload Dependence in ARDS Patients During Prone Position
Brief Title: Preload Dependence During Prone Position In ARDS Patients
Acronym: PRD-ARDS-PP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012.783
Record Dates: First submitted 2013-10-16; First posted 2013-10-18 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: ARDS PATIENTS WITH HEMODYNAMIC INSTABILITY
Keywords: ARDS - FLUID LOADING - PRELOAD DEPENDENCE
MeSH Terms: interventions — Head-Down Tilt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Procedure: Trendelenburg position

INTERVENTIONS:
Procedure: Trendelenburg position

SUMMARY:
Preload dependence assessment is difficult during prone position, and to date, no hemodynamic parameters have been validated to rationalize fluid loading in that position. This study aims to validate several hemodynamic parameters, using continuous cardiac output by pulse contour analysis and transpulmonary thermodilution.

ELIGIBILITY:
Inclusion Criteria:

* ARDS patient
* mechanically ventilated in prone position
* sedated and paralyzed
* with continuous cardiac output monitoring by transpulmonary thermodilution and pulse contour analysis
* fluid loading as indicated by attending physician

Exclusion Criteria:

* Age below 18
* no affiliation to social security
* Vena cava obstruction
* previous inclusion in protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Area under ROC curve of the variation in continuous cardiac output during Trendelenburg position, to detect preload dependence | 1 minute after Trendelenburg position onset.
  Preload dependence is assessed by the response in cardiac output to a 500 mL fluid loading, and is deemed positive if cardiac output increase by at least 15%

SECONDARY OUTCOMES:
Area under ROC curve of the variation in continuous cardiac output during end-expiratory occlusion to detect preload dependence | 15 seconds after the onset of end-expiratory occlusion
  Preload dependence is assessed by the response in cardiac output to a 500 mL fluid loading, and is deemed positive if cardiac output increase by at least 15%
Area under ROC curve of the respiratory variation in pulse pressure to detect preload dependence | 1 minute after tidal volume increase to 8 ml/kg
  Preload dependence is assessed by the response in cardiac output to a 500 mL fluid loading, and is deemed positive if cardiac output increase by at least 15%

CONTACTS AND LOCATIONS:
Overall Officials: Jean Christophe RICHARD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix Rousse, Lyon, France

REFERENCES:
- [Result] Yonis H, Bitker L, Aublanc M, Perinel Ragey S, Riad Z, Lissonde F, Louf-Durier A, Debord S, Gobert F, Tapponnier R, Guerin C, Richard JC. Change in cardiac output during Trendelenburg maneuver is a reliable predictor of fluid responsiveness in patients with acute respiratory distress syndrome in the prone position under protective ventilation. Crit Care. 2017 Dec 5;21(1):295. doi: 10.1186/s13054-017-1881-0. PMID 29208025